CLINICAL TRIAL: NCT07052487
Title: Effectiveness of Post Isometric Relaxation Technique Versus Simple Stretching Exercises for Pain and Physical Activity in Young Females With Primary Dysmenorrhea in Peshawar: A Randomized Controlled Trial
Brief Title: Effectiveness of Post Isometric Relaxation Technique Versus Simple Stretching Exercises for Pain and Physical Activity in Young Females With Primary Dysmenorrhea in Peshawar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/003
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Dysmenorrhea; Menstrual Pain
Keywords: Dysmenorrhea; Menstrual Pain; Pelvic Pain; Exercise Therapy; Physical Therapy Modalities
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: This study is a two-arm, parallel-group, randomized clinical trial with 44 participants assigned in a 1:1 ratio to either the Post-Isometric Relaxation (PIR) group or the Simple Stretching Exercises (SSE) group. Allocation will be performed centrally using a computer-generated random sequence and sealed envelopes to ensure concealment. The trial is open-label for participants, care providers, and investigators; however, outcome assessors will remain blinded to group assignments to minimize assessment bias. Primary outcomes (pain intensity via NPRS and physical activity via IPAQ) and secondary outcomes (WaLIDD score and range of motion) will be collected at baseline, week 4, and week 8 by these blinded assessors.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to each participant's group assignment. Participants, care providers, and investigators will be aware of group allocation (open-label for all other roles).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-Isometric Relaxation (PIR) (Experimental): Participants receive Post-Isometric Relaxation targeting gluteus maximus, iliopsoas, piriformis, and hamstrings. Each session begins with 10 minutes of TENS and hot-pack application, followed by for each muscle group: a 10-second isometric contraction against the therapist's counterforce, 5-second relaxation, and 30-second passive stretch, repeated three times. Sessions occur three times per week for eight weeks (24 total sessions).
  Interventions: Procedure: Post-Isometric Relaxation (PIR)
- Simple Stretching Exercises (SSE) (Active Comparator): Participants receive four basic static stretches for the gluteus maximus, iliopsoas, piriformis, and hamstrings. Each session begins with 10 minutes of TENS and hot-pack application, followed by ten repetitions of each stretch (holding each stretch for 10 seconds). Sessions occur three times per week for eight weeks (24 total sessions).
  Interventions: Procedure: Simple Stretching Exercises (SSE)

INTERVENTIONS:
Procedure: Post-Isometric Relaxation (PIR) — A manual physiotherapy technique applied to the gluteus maximus, iliopsoas, piriformis, and hamstrings. Each session begins with 10 minutes of transcutaneous electrical nerve stimulation (TENS) and moist heat (hot-pack), followed by three cycles per muscle group of: a 10-second isometric contraction against the therapist's counterforce, 5-second relaxation, and 30-second passive stretch. Sessions are delivered thrice weekly for eight weeks (24 sessions total).
  Arms: Post-Isometric Relaxation (PIR)
Procedure: Simple Stretching Exercises (SSE) — A set of four static stretches targeting the gluteus maximus, iliopsoas, piriformis, and hamstrings. Each session begins with 10 minutes of TENS and hot-pack application, followed by ten repetitions of each stretch held for 10 seconds. Sessions are delivered thrice weekly for eight weeks (24 sessions total).
  Other Names: Static Stretching Protocol
  Arms: Simple Stretching Exercises (SSE)

SUMMARY:
This randomized controlled trial will compare the effectiveness of Post-Isometric Relaxation (PIR) versus Simple Stretching Exercises (SSE), each combined with standard physiotherapy modalities, for reducing menstrual pain and improving physical activity in young unmarried women with primary dysmenorrhea. Forty-four participants will be randomly assigned (1:1) to receive either PIR or SSE three times per week for eight weeks (24 total sessions). The study will identify which non-pharmacological intervention provides superior benefits for pain relief and daily function.

DETAILED DESCRIPTION:
Primary dysmenorrhea is defined as menstrual cramps without underlying disease. This condition affects 50-90% of women of reproductive age and can significantly impair daily activities and quality of life. While pharmacologic treatments exist, non-drug interventions which include muscle energy techniques and stretching are under investigation for their safety and efficacy.

In this single-center, parallel-group randomized controlled trial, 44 unmarried female students aged 18-30 years with documented regular menstrual cycles and moderate to severe primary dysmenorrhea (WaLIDD score ≥5) will be enrolled. After baseline screening and informed consent, participants will be randomized (via OpenEpi) to one of two groups of post-isometric relaxation technique and simple stretching exercises.

Pain intensity (NPRS 0-10) and physical activity levels (IPAQ MET·min/week) will be assessed at baseline, 4 weeks, and 8 weeks by blinded assessors. Secondary measures include dysmenorrhea severity (WaLIDD questionnaire) and range of motion. Data will be analyzed with RM-ANOVA for within-group changes and independent-samples t-tests for between-group comparisons, after testing normality with Shapiro-Wilk. A p-value <0.05 denotes significance.

This trial will clarify which non-pharmacological intervention more effectively reduces menstrual pain and enhances activity, informing evidence-based physiotherapy protocols for primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-30 years.
* Self-identification as female.
* Unmarried students with regular menstrual cycles (24-35 days).
* Diagnosed primary dysmenorrhea with a WaLIDD score ≥ 5.
* Able and willing to participate in thrice-weekly physiotherapy sessions for eight weeks.
* Provide written informed consent.

Exclusion Criteria:

* Secondary dysmenorrhea (e.g., endometriosis, pelvic inflammatory disease).
* Current use of hormonal contraceptives or any medication for menstrual pain.
* History of hip or pelvic surgery in the past year.
* Acute musculoskeletal injury or chronic pain conditions unrelated to dysmenorrhea.
* Neurological disorders affecting lower-limb muscle function.
* Contraindications to TENS or heat therapy (e.g., skin lesions, implanted electronic devices).
* Pregnancy or breastfeeding.
* Participation in another interventional trial within the past three months.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants must self-identify as female.
Enrollment: 44 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Severity of Pain | Baseline, Week 4, and Week 8 (8 weeks total)
  Numeric Pain Rating Scale will be used to measure the pain intensity. Difference from baseline in average menstrual pain intensity, measured using the 11-point Numeric Pain Rating Scale (0 = no pain, 10 = worst imaginable pain). Participants rate their typical pain during the first two days of menstruation.
Physical Activity Level | Baseline, Week 4, and Week 8 (8 weeks total)
  Difference from baseline in total weekly metabolic equivalent task minutes (MET-min/week), as assessed by the short-form International Physical Activity Questionnaire.
Dysmenorrhea Severity | Baseline, Week 4, and Week 8
  Change from baseline in the Work Ability, Location, Intensity, Days of pain and Dysmenorrhea (WaLIDD) questionnaire score. The WaLIDD score ranges from 0 to 12, with higher scores indicating more severe dysmenorrhea.

SECONDARY OUTCOMES:
Compliance Rate | End of 8th week
  Percentage of prescribed sessions attended out of 24 planned sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Sheeba Orakzai, MSPT, Principal Investigator — Khyber Medical University Peshawar, Pakistan; Sibghat Ullah, MSPT, Principal Investigator — Khyber Medical University Peshawar, Pakistan
Locations (1):
- City University, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) for all enrolled subjects-including demographic variables, baseline and follow-up outcomes (NPRS scores, IPAQ MET-min/week, WaLIDD scores, hip range of motion, and session compliance)-will be made available to qualified researchers. Data will be stripped of direct identifiers in accordance with HIPAA Safe Harbor guidelines. Requests must include a methodologically sound proposal and Institutional Review Board (IRB) approval or exemption documentation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data and supporting documents will become available 12 months after publication of the primary trial results and will remain accessible for up to 5 years thereafter.
Access Criteria: Researchers must submit:
  A formal request describing the research question and analysis plan.
  Evidence of ethics approval.
  A signed data use agreement committing to protect participant confidentiality and use data only for the approved purpose.

REFERENCES:
- [Background] Kirsch E, Rahman S, Kerolus K, Hasan R, Kowalska DB, Desai A, Bergese SD. Dysmenorrhea, a Narrative Review of Therapeutic Options. J Pain Res. 2024 Aug 15;17:2657-2666. doi: 10.2147/JPR.S459584. eCollection 2024. PMID 39161419
- [Background] Ullah A, Fayyaz K, Javed U, Usman M, Malik R, Arif N, Kaleem A. Prevalence of Dysmenorrhea and Determinants of Pain Intensity Among University-Age Women. Pain Med. 2021 Dec 11;22(12):2851-2862. doi: 10.1093/pm/pnab273. PMID 34505897
- [Background] Mohamad Bakro R, Farrukh MJ, Rajagopal MS, Kristina SA, Ramatillah DL, Ming LC, Paneerselvam GS, Hadi MA. Assessment of prevalence, knowledge and health-related practices of dysmenorrhea among Malaysian women in Kuala Lumpur: a cross-sectional survey. Ann Med. 2023;55(2):2281655. doi: 10.1080/07853890.2023.2281655. Epub 2023 Nov 27. PMID 38010360
- [Background] Barbosa-Silva J, Avila MA, de Oliveira RF, Dedicacao AC, Godoy AG, Rodrigues JC, Driusso P. Prevalence, pain intensity and symptoms associated with primary dysmenorrhea: a cross-sectional study. BMC Womens Health. 2024 Feb 4;24(1):92. doi: 10.1186/s12905-023-02878-z. PMID 38311716
- [Background] Khan T, Rizvi MR, Sharma A, Ahmad F, Hasan S, Uddin S, Sidiq M, Ammari A, Iqbal A, Alghadir AH. Assessing muscle energy technique and foam roller self-myofascial release for low back pain management in two-wheeler riders. Sci Rep. 2024 May 27;14(1):12144. doi: 10.1038/s41598-024-62881-8. PMID 38802553
- [Background] Santos LBD, Barbosa IR, Dantas THM, Araujo CM, Dantas JH, Ferreira CWS, Camara SMAD, Dantas D. Prevalence of primary dysmenorrhea and associated factors in adult women. Rev Assoc Med Bras (1992). 2022 Jan;68(1):31-36. doi: 10.1590/1806-9282.20210341. PMID 35239934